CLINICAL TRIAL: NCT03735342
Title: HEARt Sounds: A Pilot Randomized Trial to Determine the Feasibility and Acceptability of Audio Recordings to Improve Discharge Communication for Cardiology Inpatients
Brief Title: HEARt Sounds: Audio Recordings to Improve Discharge Communication for Cardiology Inpatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Dartmouth College (Other)
Responsible Party: Principal Investigator, Paul J. Barr, Associate Professor, Trustees of Dartmouth College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: D18184
Record Dates: First submitted 2018-10-30; First posted 2018-11-08 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Cardiovascular Disease
Keywords: Hospital discharge; Audio-recording; Cardiology; Provider-patient communication
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Sound Recordings

STUDY DESIGN:
Who Masked: Investigator
Masking Description: To minimize selection bias, study research assistants and enrolled discharging providers are blinded to participants' (patients') study arm allocation until after participants are enrolled in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Audio Recording (Experimental): Participants receive a verbal discharge discussion with a provider, written discharge instructions and a re-playable audio recording of the discharge discussion with the discharging provider.
  Interventions: Other: Audio Recording
- Usual care (No Intervention): Participants receive a verbal discharge discussion with a provider and written discharge instructions.

INTERVENTIONS:
Other: Audio Recording — All participants will be provided with a re-playable audio recording of the discharge discussion on a portable electronic device. In addition, participants will have the option to record the discharge discussion on a personally-owned smartphone or receive access to the recording online, via the Open Recording Automated Logging System (ORALS).
  Arms: Audio Recording

SUMMARY:
Ineffective hospital discharge communication can significantly impact patient understanding, safety, and treatment adherence. This is especially true for cardiology patients, who leave the hospital with complex discharge plans, a multitude of high-risk medications, post-procedural care instructions and recommendations for drastic lifestyle changes, all delivered in a time-pressured discharge discussion. The goal of this pilot trial is to determine if it is possible to use audio recordings to supplement usual discharge communication to improve cardiology patients' ability to understand and self-manage care after leaving the hospital.

DETAILED DESCRIPTION:
The study objective is to assess the feasibility and acceptability of providing audio recorded discharge instructions to patients discharged from an inpatient cardiology service using a two-arm randomized controlled design. Specifically, this pilot study aims to: 1) Determine whether providing audio recorded discharge instructions as a supplemental discharge communication tool is feasible for cardiology providers and patients to use during the inpatient discharge discussion, 2) Determine whether it is acceptable for patients and families to use audio recorded discharge instructions after hospital discharge to self-manage care, and 3) Explore the impact of audio recording on patients' understanding of discharge instructions, ability to self-manage care and ability to adhere to prescribed medications.

On the day of discharge, enrolled patients will be randomized to a usual care arm, which includes bedside discussion and review of written discharge instructions with the discharging provider, or to an intervention arm, which includes bedside discussion and review of written discharge instructions with the discharging provider and an audio recording of that bedside discharge discussion using block randomization at the provider level. All participants randomized to the intervention arm will receive a portable, electronic recording device with audio playback that contains a recording of the bedside discharge discussion, and will also have the option to record the discharge discussion on a smartphone or receive access to the recording online, via the Open Recording Automated Logging System (ORALS). The hypothesis is providing audio recordings of discharge instructions will be feasible and acceptable to cardiology patients and providers.

One week after discharge, all enrolled patients (both arms) will be contacted via telephone to complete an interview about the use of written discharge instructions and a survey about understanding of discharge instructions, confidence and ability to self-manage care, and medication adherence. In addition, patients in the intervention arm will be interviewed about how the audio recording of the discharge discussion was used.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Cardiology inpatients
* Comfortable reading and writing in English
* Willing to have discharge conversation recorded

Exclusion Criteria:

* Patients who are unable or unwilling to provide written informed consent
* Diagnosis of dementia, schizophrenia and other psychotic disorders
* Have a substance-abuse disorder
* Severe uncorrected vision or hearing problems
* Currently living in skilled nursing facility or hospice
* Planned discharge to a structured facility (e.g., skilled nursing facility, intermediate care facility, hospice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Patient enrollment (Feasibility) | Time 1-Day of discharge, immediately post randomization
  The proportion of eligible cardiology inpatients who agreed to take part in the research.
Intervention fidelity (Feasibility) | Time 1-Day of discharge, immediately post randomization
  The proportion of cardiology inpatients in the intervention arm that received the audio recording intervention with full adherence to a pre-defined protocol fidelity checklist. Any deviations will be documented.
Patient use of intervention (Acceptability) | Time 2-One week after discharge, post randomization
  The proportion of discharged cardiology patients in the intervention arm who used the audio recording between the day of discharge and a one-week follow up telephone call initiated by the research team.

OTHER OUTCOMES:
Change in patient activation | Time 0-Day of discharge, before randomization, Time 1-Day of discharge, immediately post randomization, Time 2-One week after discharge, post randomization
  Measured using the Patient Activation Measure-13 (PAM-13). The PAM-13 is a 13-item survey that assesses a person's underlying knowledge, skills and confidence integral to managing his or her own health and healthcare. Each item is measured on a 4-point rating scale ranging from 1 (strongly disagree) to 4 (strongly agree). Scores for individual items are added to yield a sum score ranging from 0 to 100, with higher scores indicating greater self-management ability.
Change in patient health confidence | Time 0-Day of discharge, before randomization, Time 1-Day of discharge, immediately post randomization, immediately post randomization, Time 2-One week after discharge, post randomization
  The proportion of patients in the intervention arm, compared to patients in the usual care arm, who report high confidence measured using an adapted version of the Health Confidence Measure that includes three response options; "very confident", "somewhat confident" and "not confident". Response options are categorized, with "very confident" indicating high health confidence vs. "somewhat confident" and "not confident" indicating low health confidence.
Change in patient ability to understand health information | Time 0-Day of discharge, before randomization, Time 1-Day of discharge, immediately post randomization, immediately post randomization, Time 2-One week after discharge, post randomization
  The proportion of patients in the intervention arm, compared to patients in the usual care arm, who report a high ability to understand health information measured using an adapted version of the Health Confidence Measure that includes three response options; "very understandable", "somewhat understandable" and "not understandable". Response options are categorized, with "very understandable" indicating a high ability to understand health information vs. "somewhat understandable" and "not understandable" indicating a low ability to understand health information.
Change in patient general medical adherence | Time 0-Day of discharge, before randomization, Time 2-One week after discharge, post randomization
  Measured using the Medical Outcomes Study Measure of Adherence (MOS). The 5-item MOS measures general adherence to medical advice on a 6-point rating scale ranging from 1 (none of the time) to 6 (all of the time). Scores for individual items are averaged to yield a summary score ranging from 1 to 6, with higher scores indicating better adherence.
Patient assessment of discharging provider communication ability | Time 1-Day of discharge, immediately post randomization
  Measured using the Communication Assessment Tool (CAT). The 15-item CAT measures patient perceptions of physician performance in the area of interpersonal and communication skills using a 5-point rating scale ranging from 1 (poor) to 5 (excellent). The percentage of items scored as excellent is calculated as the percentage of items with a score of 5 (excellent) out of the number of items answered.
Patient adherence to medications | Time 2-One week after discharge, post randomization
  Measured using the Adherence to Refills and Medications Scale (ARMS-7). The 7-item ARMS-7 measures medication adherence and refill behaviors on a 4-point rating scale ranging from 1 (none of the time) to 4 (all of the time). Individual items are added and can be treated as a continuous measure or dichotomized as 7 or >7, with lower scores indicating better adherence.
Rate of patient-generated post-discharge phone calls | Time 2-One week after discharge, post randomization
  The number of patient-generated post-discharge phone calls to the outpatient cardiology clinic or hospital emergency telephone line between the time of discharge and the research team's post-discharge follow-up telephone interview (both arms), according to data provided by the hospital's informatics team and the electronic medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Barr, PhD, MSc, Principal Investigator — Dartmouth College; Stacey L Schott, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Derived] Schott SL, Dannenberg MD, Dodge SE, Schoonmaker JA, Caisse MM, Barr PJ, O'Malley AJ, Bruce ML. Heart sounds: a pilot randomised trial to determine the feasibility and acceptability of audio recordings to improve discharge communication for cardiology inpatients protocol. Open Heart. 2019 Jul 11;6(2):e001062. doi: 10.1136/openhrt-2019-001062. eCollection 2019. PMID 31363416